CLINICAL TRIAL: NCT06263426
Title: HOPE in Action Kidney Transplantation From Donors With HIV: Impact on Rejection and Long-Term Outcomes
Brief Title: Kidney Transplantation From Donors With HIV: Impact on Rejection and Long-Term Outcomes (Expanding HOPE Kidney)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00387066; U01AI177211 (NIH)
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV D+/R+ (Experimental): People living with HIV who receive kidneys from deceased donors with HIV
  Interventions: Other: HIV D+/R+
- HIV D-/R+ (Experimental): People living with HIV who receive kidneys from deceased donors without HIV
  Interventions: Other: HIV D-/R+

INTERVENTIONS:
Other: HIV D+/R+ — Receipt of kidney transplant from a deceased donor with HIV.
  Arms: HIV D+/R+
Other: HIV D-/R+ — Receipt of kidney transplant from a deceased donor without HIV.
  Arms: HIV D-/R+

SUMMARY:
This research is being done to better understand rejection in transplant recipients with HIV who receive kidneys from donors with vs without HIV.

DETAILED DESCRIPTION:
Previously, people with HIV in need of a transplant could only receive organs from a donor without HIV. However, in November 2013, the HIV Organ Policy Equity (HOPE) Act made it possible for people with HIV to receive organs from donors with HIV as a part of a research study.

Over the last two decades, people with HIV have received organs from donors without HIV, and in general, these recipients have done well after transplant and still maintained control of their HIV. Over the last several years, people with HIV have received organs from donors with HIV, and in general, these recipients have also done well after transplant and still maintained control of their HIV. This study will look to better understand rejection in transplant recipients with HIV (HIVR+) who receive kidneys from donors with HIV (HIVD+) vs without HIV (HIVD-).

ELIGIBILITY:
Inclusion Criteria:

* Participant meets local criteria for kidney transplant.
* Participant is able to understand and provide informed consent.
* Participant has documented HIV infection by any licensed assay or documented history of detectable HIV-1 RNA.
* Participant is ≥ 18 years old.
* HIV-1 RNA < 50 copies/mL. Viral blips between 50-400 copies will be allowed as long as there are not consecutive measurements > 200 copies/mL.
* Participant is not suffering from significant wasting (e.g. body mass index <21) thought to be related to HIV disease.

Exclusion Criteria:

* Participant has prior progressive multifocal leukoencephalopathy (PML), cryptosporidiosis of > 1 month, or primary central nervous system (CNS) lymphoma.
* Participant is pregnant or breastfeeding.
* Past or current medical problems or findings from medical history, physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of death and allograft rejection. | From date of transplant to end of year 1
  Proportion of participants who die or have graft rejection

SECONDARY OUTCOMES:
Participant survival | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Time to event (death)
Graft survival | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Time to event (graft loss)
Type and severity of graft rejection | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Based on Banff scoring criteria (kidney) for T cell- and antibody-mediated rejection (currently Banff 2019)
Time to first rejection | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Time to event (first rejection)
Rate of rejection events over time | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Count of rejection events
Graft function over time measured by eGFR trajectory | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Estimated glomerular filtration rate, calculated centrally based on local testing results
Incidence of HIV viremia post-transplant | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Cumulative incidence of HIV viremia based on local testing
Incidence of new antiretroviral drug resistance and/or X4 tropic virus posttransplant | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Cumulative incidence of new resistance and/or X4 tropic virus based on local testing
Incidence of bacterial, fungal, viral, and other opportunistic infections posttransplant | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Cumulative incidence of infections
Incidence of surgical and vascular transplant complications post-transplant | In the first year post-transplant
  Cumulative incidence of complications
Incidence and causes of chronic kidney disease post-transplant | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Cumulative incidence of chronic kidney disease (eGFR<60 for more than 3 months)
Incidence of post-transplant malignancies | From transplant through end of follow up (at least 1 year, up to 4 years post-transplant)
  Cumulative incidence of malignancies
Incidence of de novo donor specific antibody (DSA) | At month 12 post-transplant
  Based on central testing

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Columbia University, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania